CLINICAL TRIAL: NCT07347743
Title: Double-blind, Randomized Placebo-controlled Trial for the Preventive Effect of Limosilactobacillus Reuteri (L. Reuteri) on Excessive Crying and Colic in Healthy Infants.
Brief Title: Preventive Effect of a Dietary Supplement With Two Probiotic Limosilactobacillus Reuteri Strains on Excessive Crying and Colic in Healthy Newborns.
Acronym: ProtectPrevent
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: BioGaia AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Prot-Prev
Record Dates: First submitted 2025-12-09; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-10

CONDITIONS: Colic; Healthy Infants; Eczema Atopic Dermatitis
Keywords: Preventive effect; Limosilactobacillus reuteri; L. reuteri; crying; colic; healthy infants; newborns; DSM 17938; BG-R46™
MeSH Terms: conditions — Colic; Crying

STUDY DESIGN:
Intervention Model Description: Prospective, double-blind, parallel, randomized, placebo-controlled superiority trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): The control groups gets no Limosilactobacillus reuteri
  Interventions: Dietary Supplement: Placebo
- Intervention group (Experimental): The intervention group gets the two probiotic Limosilactobacillus reuteri strains
  Interventions: Dietary Supplement: Two probiotic Limosilactobacillus reuteri strains

INTERVENTIONS:
Dietary Supplement: Two probiotic Limosilactobacillus reuteri strains — Each participant in this intervention group gets 5 drops per day, containing the two probiotic Limosilactobacillus reuteri strains (DSM 17938 and BG-R46™) and 400 IU of Vitamin D
  Arms: Intervention group
Dietary Supplement: Placebo — Each participant in this intervention group gets 5 drops per day, containing only 400 IU of Vitamin D.
  Arms: Control group

SUMMARY:
This study aims to demonstrate that a dietary supplement, which contains two strains (DSM 17938 and BG-R46TM) of the probiotic L. reuteri is safe, well tolerated and able to reduce the incidence of colic and excessive crying/fussiness in healthy infants. Additionally, the study aims to investigate if children with this probiotic supplement have better stool characteristics and a more beneficial composition of the fecal and skin flora than children given a placebo during the first 3 months of life.

DETAILED DESCRIPTION:
This study is a double-blind, randomized, placebo-controlled trial conducted at UZ Brussel to evaluate the safety and preventive efficacy of a dietary supplement containing two probiotic strains, Limosilactobacillus reuteri DSM 17938 and BG-R46™, on excessive crying and the development of infantile colic in healthy newborns.

Recent systematic reviews and meta-analyses have shown that supplementation with L. reuteri DSM 17938 significantly reduces crying and fussing time in infants. A novel formulation combining DSM 17938 with BG-R46™ was developed to achieve a potentially enhanced effect on infant distress symptoms. This study investigates whether early supplementation, initiated within the first week of life, is safe and effective during the first three months of life.

Healthy, full-term infants (≥37 weeks' gestation) aged 1-14 days at inclusion are eligible. Participants are randomized to receive either placebo plus vitamin D (400 IU) or L. reuteri DSM 17938 and BG-R46™ plus vitamin D (400 IU) for a maximum of 98 days, until approximately 3 months of age.

Study visits include a baseline visit (day 1-14), a midway visit at 6 weeks, an end-of-intervention visit at 3 months, and a long-term follow-up at 1 year. Additional telephone contacts are triggered by infant day diaries.

The primary outcomes are peak crying and fussing time at 6 weeks of age and the occurrence of infantile colic during the first 3 months of life. Secondary outcomes include infant quality of life (ITQOL™), parental stress, parental satisfaction, crying and fussiness patterns, and the presence of atopic dermatitis. Exploratory outcomes assess changes in the intestinal microbiome, stool characteristics, biomarkers, growth, and allergy-related parameters.

The primary hypothesis is that daily supplementation with L. reuteri DSM 17938 and BG-R46™ reduces the incidence of infantile colic and peak crying time at 6 weeks. Secondary hypotheses propose microbiome modulation leading to reduced distress, improved infant quality of life, and lower parental stress.

ELIGIBILITY:
Inclusion Criteria:

1. Infant is born at the maternity ward of UZ Brussel with a gestational age of ≥37 weeks.
2. Infant is healthy at the time of pre-examination.
3. Infant is aged between 1 and 14 days old at the time of inclusion.
4. Legal guardian(s) are able and willing to follow the study instructions
5. Infant is suitable for participation in the study according to the investigator/ study personnel
6. Legal guardian(s) willing to refrain products containing probiotics for their infant, from baseline (visit 1) throughout the study period (visit 3).
7. Informed written consent given by parent / legal guardian

Exclusion Criteria:

1. No legal guardian's command of any local language
2. Infant with a major congenital anomaly (i.e. anal atresia, trisomy 21) or suspicion of any chronic disorder or disease (i.e. Hirschsprung's disease, metabolic disorder)
3. Infant is suffering from congenital or acquired immunodeficiency
4. Infant is suffering from an infection at the time of pre-examination or previous 7 days
5. Infant is admitted post-partum to the neonatal intensive care unit
6. Infant is not suitable for participation in the study according to the study personnel´s opinion

Ages: 1 Day to 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 768 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-05 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Peak measured crying time | 6 weeks
  Peak measured crying time at 6 (±1) weeks according to the prospectively kept baby day diary
The occurrence of infant colic at any time in the first 3 months of life. | 3 months
  The criteria for infant colic are:
  * Recurrent and prolonged periods of infant crying, fussing, or irritability reported by caregivers that occur without obvious cause and cannot be prevented or resolved by caregivers. Fussing refers to intermittent distressed vocalization and refers to behavior that is not quite crying but not awake and content either.
  * Caregiver reports infant has cried or fussed for 3 or more hours/day during 3 or more days in a given week.
  * Total 24-hour crying plus fussing in the selected group of infants is confirmed to be 3 hours or more when measured by at least one, prospectively kept, 24-hour behavior diary.

SECONDARY OUTCOMES:
Peak measured fussiness time | 6 weeks
  Peak measured fussiness time at the age of 6 (±1) weeks according to the prospectively kept baby day diary.
Overall crying and/or fussiness time | 3 months
  Overall (estimated + measured) crying and/or fussiness time in the first 3 months (±1 week) of life.
Overall unconsolable crying time | 3 months
  Overall measured and/or estimated unconsolable crying time in the first 3 months (±1 week) of life
Parental stress | 3 months
  Parental stress as measured by the Parental Stress Scale (PSS) at 6 (±1) weeks and 3 months (±1 week) of both (if applicable) caregivers. Parents can indicate the degree to which they agree or disagree with the statements in this questionnaire, ranging from strongly disagree (1 point) to strongly agree (5 points). Total scores range from 18 points (low score signify a low level of stress) to 90 points (high score signify a high level of stress).
Quality of Life score | 12 months
  Infant and toddler quality of life questionnaire(ITQOL™) at 3 months (±1 week) and of 12 months (±2 weeks) age. ITQOL is scored on a scale from 0 to 100, where higher scores mean better health/quality of life.
Parental satisfaction | 3 months
  Parental satisfaction scale measured by a 5-point Likert scale at 6 (±1) weeks and 3 months (±1 week). A scale where parents indicate how satisfied they are with their baby's current level of crying and fussing, with a minimum score of 2 and maximum score of 10. Parents who are very dissatisfied have a low score, while parents who are very satisfied have a high score.
Atopic dermatitis | 12 months
  Presence and degree of atopic dermatitis (AD, measured via SCORAD) at 3 months (±1 week) and 12 months (±2 weeks) of age. The score ranges from 0 to 103 and is used to determine the stages of AD severity. Where a score lower than 25 is seen as mild state, 25-50 is a moderate state and >50 is a severe state.

OTHER OUTCOMES:
Stool consistency | 3 months
  Assessed by the parents in a continuous daily bowel diary over the study period using the Brussels infant and toddler stool scale (BITSS). BITSS was validated as a reliable instrument to assess stools of non-toilet trained children There are 4 possible answers: A: Hard stool, B: Formed stool, C: Loose Stool and D: Watery stool, based on pictures.
Stool frequency | 3 months
  assessed by the parents and day care centers in a continuous daily bowel diary over the study period using the BITSS
Fecal calprotectine levels | 3 months
  Fecal calprotectin at 6 (±1) weeks and 3 months (±1 week) of age
Saliva melatonin levels | 3 months
  Morning saliva melatonin level at 6 (±1) weeks and 3 months (±1 week) of age
Safety outcomes - Adverse events | 3 months
  Number of (serious) adverse events throughout the study period. Parents are asked to provide detailed information on any adverse events their child may experience during the study. For each event, the diagnosis, sign, or symptom is written down, as well as the date the event started and ended. Parents should also describe the severity of the event, rating it as mild, moderate, or severe, and provide their assessment of its relationship to the study product, categorizing it as unrelated, unlikely, probable, or related. Moreover the outcome of the event should be specified, such as fatal, not resolved, resolved, resolved with sequelae, resolving, or unknown. Lastly, parents should report any actions taken regarding the study product, including whether the dose was unchanged, reduced, increased, temporarily suspended, or definitively withdrawn, or if there was any concomitant medication given to the child or no action was required.
Weight | 3 months
  Weight for age z score at each study visit
Stool pH | 3 months
  Stool pH at 6 (±1) weeks and 3 months (±1 week)
Short Chain Fatty Acids (SCFA) | 3 months
  SCFA analysis at 6 (±1) weeks and 3 months (±1 week) of age. Concentrations of both straight-chain SCFA as branched-chain SCFA will be measured to be associated with the health status of the gut microbiota.
Skin microbiome | 12 months
  16S ribosomal RNA (rRNA) gene amplicon sequencing of skin microbiome (or shotgun metagenomics sequencing if the budget allows for this) at 6 weeks, 3 months and 12 months. To gain insight into the quantitative and qualitative abundance of microbial composition and diversity
Stool microbiome | 3 months
  16S ribosomal RNA (rRNA) gene amplicon sequencing of stool microbiome (or shotgun metagenomics sequencing if the budget allows for this) at 6 weeks, 3 months. To gain insight into the quantitative and qualitative abundance of microbial composition and diversity
Height | 3 months
  Height for age Z-score at each study visit
Weight for height | 3 months
  Weight for height z score at each study visit

CONTACTS AND LOCATIONS:
Overall Officials: Koen Huysentruyt, Pediatric Gastroenterologist, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- Universitair Ziekenhuis Brussel, Jette, Brussels Capital, Belgium